CLINICAL TRIAL: NCT06010160
Title: A Hybrid Implementation-Effectiveness Trial of Game Changers for Cervical Cancer Prevention in Uganda
Brief Title: Game Changers for Cervical Cancer Prevention
Acronym: GC-CCP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: Makerere University (Other); African Palliative Care Association (Unknown); Rays of Hope Hospice Jinja (Unknown); Indiana University, Bloomington (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023-N0111
Record Dates: First submitted 2023-08-17; First posted 2023-08-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: Individual randomization to one of two parallel groups, the intervention or usual care (no intervention) control group
Who Masked: Outcomes Assessor
Masking Description: The assessment interviewer will be blinded to study arm allocation of the participants at baseline only
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advocacy Training Intervention (Experimental): 6 weekly group sessions of advocacy training for cervical cancer screening
  Interventions: Behavioral: Game Changers for Cervical Cancer Prevention
- Usual care control (No Intervention): usual care (no intervention); control participants will be offered the chance to receive the intervention at the conclusion of month 12 follow-up data collection

INTERVENTIONS:
Behavioral: Game Changers for Cervical Cancer Prevention — The peer advocacy training sessions focus on reduction of internalized stigma, disclosure decision making, education on cervical cancer facts and myths, and building skills for cervical cancer prevention advocacy.
  Other Names: GC-CCP
  Arms: Advocacy Training Intervention

SUMMARY:
This randomized controlled trial will evaluate Game Changers for Cervical Cancer Prevention (GC-CCP) for increasing cervical cancer (CC) screening advocacy among intervention recipients (index participants) towards female social network members, and uptake of CC screening among enrolled female social network members (alter participants) who have not previously been screened. The main research questions are:

1. Is the GC-CCP network-based peer advocacy intervention superior to usual care (no intervention) in improving uptake of CC screening among alter participants, across urban/rural and public/private clinics?
2. What are the mediators and moderators (among index, alter and network characteristics) of intervention effects on (a) alter CC screening; and (b) engagement in CC prevention advocacy among index participants?

DETAILED DESCRIPTION:
This randomized controlled trial will evaluate Game Changers for Cervical Cancer Prevention (GC-CCP) for increasing cervical cancer (CC) screening among previously unscreened social network members. The trial will be conducted at 4 study clinics [2 public, 2 private-not-for-profit (PNFP), one each in an urban and rural location]. At each clinic, 40 women screened for CC in the past year will be enrolled in the RCT as index participants (n=160 index) and randomized to the intervention (in two groups of 10) or wait-list control. The intervention will consist of 6 weekly group sessions that focus on CC stigma reduction, sharing of CC screening experience with others, knowledge of CC facts and myths, and skills building for engagement in CC prevention advocacy with female social network members (1st degree alters). Each index will recruit up to three alters (n~440 1st degree alters) at baseline who have not screened for CC; these index and alter participants will be followed up at months 6 and 12. At month 6, half of the 1st degree alters will be asked to recruit up to female social network members (2nd degree alters) whom they have engaged in CC screening advocacy with; these 2nd degree alters will receive a single phone-based brief interview; at month 12, the other half of the 1st degree alters will be asked to recruit up to two 2nd degree alters for the same purpose.

ELIGIBILITY:
Inclusion Criteria:

* screened for cervical cancer in the past year (index participants only)
* has shared cervical cancer screening experience with at least one adult female social network member whom is believed to not have been screening for cervical cancer; or she reports that there is at least one female social network member who has not screened and she would feel comfortable disclosing her personal screening experience to her (index participants only)
* is a member of social network of enrolled participant (social network member participants only)

Exclusion Criteria:

* advanced stage cervical cancer (index participants only)
* screened for cervical cancer in the past (1st degree social network member participants only)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Number of alter participants that has received cervical cancer screening | past 6 months
  Receipt of screening via visual inspection of cervix with acetic acid (VIA), among enrolled alter participants

SECONDARY OUTCOMES:
Mean score on cervical cancer prevention advocacy scale | past 6 months
  6-item Self-reported scale of engagement in CC prevention advocacy (each item using a 1-5 scale), among index participants; higher scores reflect greater advocacy

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Wagner, PhD, Principal Investigator — RAND
Locations (1):
- Makerere University School of Public Health, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
A de-identified dataset will be made available upon review of requests from outside researchers
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Following publication of primary results of the study, for 3 years

REFERENCES:
- [Derived] Wagner GJ, Bogart LM, Matovu JKB, Gwokyalya V, Beyeza-Kashesya J, Ober A, Green HD, Nakami S, Juncker M, Namisango E, Luyirika E, McBain RK, Bouskill K, Wanyenze RK. Study protocol for a hybrid implementation-effectiveness trial of Game Changers for Cervical Cancer Prevention in Uganda. PLoS One. 2025 Jan 24;20(1):e0317491. doi: 10.1371/journal.pone.0317491. eCollection 2025. PMID 39854403